CLINICAL TRIAL: NCT03882125
Title: Mindfulness-Based Relapse Prevention for Methadone Maintenance: A Feasibility Trial
Brief Title: Mindfulness-Based Relapse Prevention for Methadone Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific University (Other)
Responsible Party: Principal Investigator, Sarah Bowen, Assistant Professor, Pacific University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBRP for MMT
Record Dates: First submitted 2017-04-03; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Substance-Related Disorders
Keywords: mindfulness; methadone maintenance; relapse prevention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness (Experimental): Assigned to a 6-week mindfulness-based relapse prevention course
  Interventions: Behavioral: Mindfulness-based relapse prevention

INTERVENTIONS:
Behavioral: Mindfulness-based relapse prevention — Psychosocial intervention integrating mindfulness practice and cognitive behavioral relapse prevention approaches

SUMMARY:
The current study was designed to inform protocol adaptation, and to evaluate the feasibility, acceptability, and preliminary efficacy of a mindfulness-based intervention for methadone maintenance clients. Adults (N=15) were recruited from a methadone clinic to participate in a 6-week mindfulness course. Indices of feasibility, including recruitment, retention, data from focus groups and course satisfaction surveys, supported feasibility of the intervention. Outcome measures were self-report, and included depression, craving, PTSD symptoms, and experiential avoidance, and were assessed at baseline, postcourse, and 1-month follow-up. Data were analyzed using qualitative and quantitative approaches. Mean scores on all primary outcomes changed in the expected direction at both postcourse and 1-month follow-up assessment, although only depression and experiential avoidance reached significance. Results support feasibility and acceptability, and provide preliminary data on outcomes for future trials of mindfulness-based approaches within this client population.

DETAILED DESCRIPTION:
As rates of opiate misuse rise in the United States, there areso do significant associated health, and financial consequences to afflicted individuals, their families, and society at large. Methadone Maintenance Therapy (MMT) is one evidence-based approach to treating individuals with opiate addiction, yet supplemental psychosocial treatment to support this approach is lacking. Mindfulness-Based Relapse Prevention (MBRP) has shown to be efficacious in various substance use populations, but has yet to be assessed with MMT clients. The current study was designed to inform protocol adaptation for to MMT clients, and to evaluate the feasibility, acceptability, and preliminary efficacy of a MBRP for this population. The sample consisted of adults (N=15) recruited from a methadone clinic to participate in a 6-week MBRP course. Indices of feasibility, including recruitment, retention, data from focus groups and course satisfaction surveys, supported feasibility of the intervention. Outcome measures were self-report, and included self-compassion, depression, craving, PTSD symptoms, and experiential avoidance, and were assessed at baseline, postcourse, and 1-month follow-up. Data were analyzed using qualitative and quantitative approaches. Mean scores on all primary outcomes changed in the expected direction at both postcourse and 1-month follow-up assessment, although only depression and experiential avoidance reached significance. Results from this initial pilot support feasibility and acceptability, and provide preliminary data on outcomes for future trials of mindfulness-based approaches within the MMT community.

ELIGIBILITY:
Inclusion Criteria:

* Clearance from clinic staff
* Currently enrolled in a methadone maintenance program
* Agree to complete assessment questionnaires and attend treatment sessions
* Fluent in English

Exclusion Criteria:

* Indication of active psychosis
* Participation in past mindfulness-based relapse prevention group

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-02-15 (Actual); Primary Completion 2015-06-27 (Actual); Study Completion 2015-06-27 (Actual)

PRIMARY OUTCOMES:
Acceptability - Satisfaction with the Course | post course (6 weeks)
  Satisfaction with the course will be assessed using the Overall Course Satisfaction Survey, items #1-4 (Bowen, Chawla, & Marlatt, 2010). This is a self-report questionnaire, the first 4 items of which are open-ended questions assessing satisfaction with the course, barriers to learning, and perceived helpfulness.
Acceptability - Enactment of Learned Skills | post course (6 weeks)
  Enactment will be assessed using the Overall Course Satisfaction Survey, items #5-7 (Bowen, Chawla, & Marlatt, 2010). This is a self-report questionnaire, the last 3 questions of which are 10-point Likert-type items, and assess importance of skills and likelihood of implementing them into daily life after the course ends. Higher scores indicate higher perceived importance and likelihood.

SECONDARY OUTCOMES:
Depression | 1 month
  Depression symptoms will be assessed using the Beck Depression Inventory-II, a 21-item self report measure. Items are summed for a total score ranging from 0-63. A score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Anxiety | 1 month
  Anxiety symptoms will be assessed using the Beck Anxiety Inventory, a 21-item self report measure. Items are summed for a total score that can range between 0 and 63 points. A total score of 0 - 7 is interpreted as a Minimal anxiety, 8 - 15 as Mild, 16 - 25 as Moderate, and 26 - 63 as Severe.
Craving | 1 month
  Craving for substances will be assessed using the Penn Alcohol Craving Scale, a five-item Likert-scaled measure assessing frequency, intensity, duration, and overall levels of craving, adapted to include both alcohol and drugs. Each question is scaled from 0 to 6. Sum scores range from 0-30, with greater scores indicating higher craving.
Trauma symptoms | 1 month
  PTSD symptoms will be assessed using the Post-Traumatic Stress Disorder Checklist-Civilian (PCL-C), which measures presence and severity of trauma symptoms using 16-item Likert-scaled questionnaire.
Experiential avoidance | 1 month
  The Acceptance and Action Questionnaire (AAQ) is a widely used measure of experiential avoidance and psychological inflexibility consisting of nine Likert-scaled items, answer options ranging from 1 (never true) to 7 (always true). High scores reflect greater experiential avoidance and immobility, while low scores reflect greater acceptance and action.

IPD SHARING:
Plan to Share IPD: Undecided